CLINICAL TRIAL: NCT01472120
Title: The Relationship of Adiponectin With Circulating Macrophage Phenotypes in Non-alcoholic Fatty Liver Disease
Brief Title: Adiponectin and Circulating Macrophage Phenotypes in Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Halil Genc, Gulhane School of Medicine, Gulhane School of Medicine
Other Study IDs: NASH-macrophage
Record Dates: First submitted 2011-08-11; First posted 2011-11-16 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-08

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- P and C: P: NAFLD patients
  C: Healthy controls

SUMMARY:
In peripheral blood; monocytes and macrophages are found in two phenotype; proinflammatory M1 and anti-inflammatory M2 phenotypes. M2 form is converted (or polarized) to M1 phenotype in various metabolic disorders such as obesity and type 2 diabetes mellitus.

DETAILED DESCRIPTION:
In peripheral blood; monocytes and macrophages are found in two phenotype; proinflammatory M1 and anti-inflammatory M2 phenotypes.

M2 form is converted (or polarized) to M1 phenotype in various metabolic disorders such as obesity and type 2 diabetes mellitus. In addition, these forms also are related to insulin resistance and inflammation in adipose tissue.

Today, there is no study that investigate the role of adiponectin an anti-inflammatory adipokine, on macrophage polarization in non-alcoholic fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Persistently (at least 6 months) elevated aminotransferases
* Ultrasonographic presence of bright liver without any other liver or biliary tract disease
* Liver histology compatible with a diagnosis of NASH or SS

Exclusion Criteria:

* A history of alcohol consumption >40 g/wk, as assessed by a detailed interview extended to family members
* Morbid obesity [body mass index (BMI) ≥40 kg/m2], hypertension
* Positive blood markers of viral, autoimmune, or celiac disease
* Abnormal copper metabolism or thyroid function tests
* A diagnosis of T2DM and systemic arterial hypertension
* Total cholesterol (TC) ≥250 mg/dL, triglycerides (TG) ≥400 mg/dL, exposure to occupational hepatotoxins or drugs known to affect glucose and lipid metabolism

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A sample of male outpatients with histologically proven NAFLD, who attended the outpatient clinic of the Gastroenterology Department, Gulhane School of Medicine, Ankara, Turkey
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-09 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
For laboratory analyses, the collection of all blood samples from the study participants. | Collection of blood samples in one year and analyses of data in 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: halil genc, MD, Principal Investigator — Gulhane Medical School
Locations (1):
- Gastroenterology Department, Gulhane School of Medicine, Ankara, Turkey (Türkiye)